CLINICAL TRIAL: NCT00280371
Title: A 12-week Double-Blind, Parallel-Group, Placebo- and Active- Controlled Trial to Evaluate the Efficacy and Safety of Formoterol Fumarate Inhalation Solution 20 Mcg/0.5 mL Delivered by OMRON MicroAir NE-U22V Nebulizer in the Treatment of Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Trial to Evaluate the Efficacy and Safety of Formoterol Fumarate 20 Mcg/0.5 mL in the Treatment of Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Director, Clinical Affairs, Dey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201-069
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2008-02

CONDITIONS: COPD
Keywords: COPD; Chronic Obstructive Pulmonary Disease; formoterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

INTERVENTIONS:
Drug: Formoterol Fumarate

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the investigational drug in comparison with a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of COPD
* Current or prior history of cigarette smoking

Exclusion Criteria:

* Medical diagnosis of asthma
* Chest X-ray diagnostic of significant disease other than COPD
* Significant condition or disease other than COPD

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345
Dates: Start 2006-01; Primary Completion 2006-07 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Measure of lung function

SECONDARY OUTCOMES:
Change in lung function, as well as vital signs
Physical Exam results, adverse event reporting, etc

CONTACTS AND LOCATIONS:
Locations (50):
- United States (50):
  - Research Site, Jasper, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Buena Park, California
  - Research Site, Costa Mesa, California
  - Research Site, Huntington Beach, California
  - Research Site, Long Beach, California
  - Research Site, San Diego, California
  - Research Site, Stockton, California
  - Research Site, Walnut Creek, California
  - Research Site, Denver, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Clearwater, Florida
  - Research Site, DeLand, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Hines, Illinois
  - Research Site, Normal, Illinois
  - Research Site, Overland Park, Kansas
  - Research Site, Shawnee Mission, Kansas
  - Research Site, Topeka, Kansas
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Henderson, Nevada
  - Research Site, Summit, New Jersey
  - Research Site, Camillus, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Elizabeth City, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Upland, Pennsylvania
  - Research Site, Cranston, Rhode Island
  - Research Site, Spartanburg, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Waco, Texas
  - Research Site, South Burlington, Vermont
  - Research Site, Abingdon, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin